CLINICAL TRIAL: NCT05534399
Title: Assessment of the Interest of a Peri-operative Antibiotic Strategy Applied to Patients With Asymptomatic Bacteriuria Undergoing Intra-vesical Botulinum Toxin A Injections
Brief Title: Antibiotic Strategy and Asymptomatic Bacteriuria in the Context of Intra-vesical Botulinum Toxin A Injections.
Acronym: ANTIBIOBONTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020_03; 2020-A03361-38 (Other: ID-RCB number,ANSM); PHRC-19-0218 (Other: DGOS number, PHRC-N)
Record Dates: First submitted 2022-06-07; First posted 2022-09-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Urinary Tract Disease
Keywords: Neurogenic lower urinary tract dysfunction; Clean Intermittent Self Catheterization; Asymptomatic bacteriuria; Botulinum toxin A; Sparing antibiotic strategy; Safety
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sparing antibiotic strategy (Experimental): No antibiotic therapy will be administered during the peri-operative period
  Interventions: Procedure: Intra-vesical BoNTA injections
- Peri-operative antibiotic strategy (Sham Comparator): Recommendations - An antibiotic therapy will be administered during the peri-operative period.
  The antibiotic will be selected according to the type of bacteria isolated and the antibiotic susceptibility testing, and started two days before and pursued until two days following intra-vesical BoNTA injections
  Interventions: Procedure: Intra-vesical BoNTA injections

INTERVENTIONS:
Procedure: Intra-vesical BoNTA injections — Intra-vesical BoNTA injections will be performed according to the protocol currently applied by the department.
  They will be performed in the operating room or in the outpatient clinic under strict asepsis, including the wearing of sterile gloves by the surgeon associated with an antiseptic brushing of the patient and the establishment of sterile fields.
  A rigid or a flexible cystoscope will be used.
  After the introduction of the cystoscope under visual control, complete bladder emptying will be performed. The bladder will be filled again, slowly and at low pressure to allow the bladder mucosa to expand.
  BoNTA (BOTOX® 200 U) will be diluted as follows: BOTOX® 200 U: in 30 mL of saline solution
  The solution obtained will be injected all along the bladder wall, sparing the trigone in 20 (BOTOX® 200 U) points using a Bonee®-type needle.
  A complete bladder emptying will be performed at the end of the procedure.

SUMMARY:
The study aims to demonstrate that the "thrifty antibiotic strategy" applied to MS or SCI patients with asymptomatic bacteriuria prior to BoNTA intravesical injections does not increase the rate of symptomatic post-injection UTIs compared to the current peri-operative antibiotic strategy.

Patients included in the study will be randomized in two balanced-parallel groups, 4 days (+/- 2 days) before intra-vesical BoNTA injections.

Group 1: Experimental group: "Sparing antibiotic strategy" No antibiotic therapy will be administered during the peri-operative period.

Group 2: Control group: Recommendations - Peri-operative antibiotic strategy An antibiotic therapy will be administered during the peri-operative period. The antibiotic will be selected according to the type of bacteria isolated and the antibiotic susceptibility testing, and started two days before and pursued until two days following intra-vesical BoNTA injections.

The main objective is to demonstrate the non-inferiority of "antibiotic saving strategy" compared to peri-operative antibiotic strategy (current recommendations) for occurrence of symptomatic UTI after intra-vesical BoNTA injections in the management of asymptomatic bacteriuria (AB) among multiple sclerosis (MS) and spinal cord injured (SCI) patients undergoing clean intermittent self-catheterization (CISC).

ELIGIBILITY:
Inclusion Criteria:

* MS or SCI (traumatic or non-traumatic)
* Refractory OAB and/or DO (failure, intolerance or contra-indication to anti-muscarinic therapy)
* Treated with intra-vesical botulinum toxin A injections having proved efficacy
* CISC as the exclusive bladder management
* AB on pre-operative urine analysis (performed 10 days (+/- 2 days) before intra-vesical BoNTA injections)
* Exclusion of morphologic urinary tract abnormalities considered as a risk factor for recurrent symptomatic UTI.

Exclusion Criteria:

* Having already participated to the study
* Augmentation cystoplasty
* Bladder compliance disorders (<20 mL/cmH2O)
* Ongoing cyclic antibiotic therapy
* Ongoing corticosteroid therapy
* Modification of immunosuppressive or immunomodulatory therapy in the 3 months before inclusion (MS patients)
* Antibiotic therapy in the month before inclusion
* Surgical procedure in the 3 months before and the 6 weeks following inclusion
* Symptomatic UTI at the time of inclusion
* Associated neurologic disease
* Pregnancy or breast feeding
* Individuals especially in need of protection
* No informed consent
* Patients incapable to follow the trial, e.g. because of language problems, psychiatric disorders, dementia and so on
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with symptomatic UTI occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Symptomatic UTI will be defined according to the National Institute on Disability and Rehabilitation Research (NIDRR, 1992) as a significant bacteriuria with tissue invasion and resultant tissue response with signs and/or symptoms of UTI

SECONDARY OUTCOMES:
Rate of patients with febrile symptomatic UTI occurring within the 6 weeks following BoNTA injections.occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Symptomatic UTI will be defined according to the National Institute on Disability and Rehabilitation Research (NIDRR, 1992) as a significant bacteriuria with tissue invasion and resultant tissue response with signs and/or symptoms of UTI
Rate of patients with non-febrile symptomatic UTI occurring within the 6 weeks following BoNTA injections | During the 6 weeks following the injections
  Symptomatic UTI will be defined according to the National Institute on Disability and Rehabilitation Research (NIDRR, 1992) as a significant bacteriuria with tissue invasion and resultant tissue response with signs and/or symptoms of UTI
Rate of patients with symptomatic UTI within the 6 weeks following BoNTA injections finally needing the administration of an antibiotic therapy. | During the 6 weeks following the injections
  Symptomatic UTI will be defined according to the National Institute on Disability and Rehabilitation Research (NIDRR, 1992) as a significant bacteriuria with tissue invasion and resultant tissue response with signs and/or symptoms of UTI
Rate of patients with complication (other than symptomatic UTI) related to* BoNTA injections occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Any complication leading to an admission in an emergency unit : macroscopic hematuria persisting for more than 48 hours after injections, painful catheterization lasting more than 48 hours after intra-vesical BoNTA injections, pseudo-botulism, botulism.
Rate of patients with complication not related to** BoNTA injections occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Any complication not listed in the complications "related to" the injections
Rate of patients with admission to an emergency unit related to* BoNTA injections occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Any complication leading to an admission in an emergency unit : macroscopic hematuria persisting for more than 48 hours after injections, painful catheterization lasting more than 48 hours after intra-vesical BoNTA injections, pseudo-botulism, botulism.
Rate of patients with admission to an emergency unit not related** to BoNTA occurring within the 6 weeks following the injections | During the 6 weeks following the injections
  Any complication not listed in the complications "related to" the injections.
Rate of patients with admission in a non-scheduled hospitalization related to* BoNTA injections occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Any complication leading to an admission in an emergency unit : macroscopic hematuria persisting for more than 48 hours after injections, painful catheterization lasting more than 48 hours after intra-vesical BoNTA injections, pseudo-botulism, botulism.
Rate of patients with admission in a non-scheduled hospitalization not related to* BoNTA injections occurring within the 6 weeks following the injections. | During the 6 weeks following the injections
  Any complication not listed in the complications "related to" the injections.
Maximal cystometric capacity (MCC) | 6 weeks after BoNTA injections.
  Maximal cystometric capacity (MCC) measured during the urodynamic multichannel study
Rate of patients with detrusor overactivity (non-voiding detrusor contractions during feeling phase) | 6 weeks after BoNTA injections.
  Detrusor overactivity measured during the urodynamic multichannel study
Number of CISC per day | 6 weeks after BoNTA injections.
  Number of CISC measured on a 3-day bladder diary
Number of urgency episodes per day | 6 weeks after BoNTA injections.
  Number of urgency episodes measured on a 3-day bladder diary
Number of urinary incontinence episodes per day | 6 weeks after BoNTA injections.
  Number of urinary incontinence episodes measured on a 3-day bladder diary
Functional bladder capacity | 6 weeks after BoNTA injections.
  Functional bladder capacity measured on a 3-day bladder diary
Identify risk factors of in-hospital postoperative symptomatic UTI | 6 weeks after BoNTA injections.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier BIARDEAU, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

REFERENCES:
- [Background] Leitner L, Sammer U, Walter M, Knupfer SC, Schneider MP, Seifert B, Tornic J, Mehnert U, Kessler TM. Antibiotic prophylaxis may not be necessary in patients with asymptomatic bacteriuria undergoing intradetrusor onabotulinumtoxinA injections for neurogenic detrusor overactivity. Sci Rep. 2016 Sep 12;6:33197. doi: 10.1038/srep33197. PMID 27616488
- [Background] Weglinski L, Rouzaud C, Even A, Bouchand F, Davido B, Duran C, Salomon J, Perronne C, Denys P, Chartier-Kastler E, Dinh A. Prospective evaluation of antibiotic treatment for urological procedure in patients presenting with neurogenic bladder. Med Mal Infect. 2016 Sep;46(6):300-7. doi: 10.1016/j.medmal.2016.04.001. Epub 2016 May 27. PMID 27241225
- [Background] Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. BMJ. 2010 May 18;340:c2096. doi: 10.1136/bmj.c2096. PMID 20483949
- [Background] Kang MS, Lee BS, Lee HJ, Hwang SW, Han ZA. Prevalence of and Risk Factors for Multidrug-Resistant Bacteria in Urine Cultures of Spinal Cord Injury Patients. Ann Rehabil Med. 2015 Oct;39(5):686-95. doi: 10.5535/arm.2015.39.5.686. Epub 2015 Oct 26. PMID 26605166
- [Background] Hansson S, Jodal U, Lincoln K, Svanborg-Eden C. Untreated asymptomatic bacteriuria in girls: II--Effect of phenoxymethylpenicillin and erythromycin given for intercurrent infections. BMJ. 1989 Apr 1;298(6677):856-9. doi: 10.1136/bmj.298.6677.856. PMID 2497823
- [Background] Cai T, Mazzoli S, Mondaini N, Meacci F, Nesi G, D'Elia C, Malossini G, Boddi V, Bartoletti R. The role of asymptomatic bacteriuria in young women with recurrent urinary tract infections: to treat or not to treat? Clin Infect Dis. 2012 Sep;55(6):771-7. doi: 10.1093/cid/cis534. Epub 2012 Jun 7. PMID 22677710